CLINICAL TRIAL: NCT04680702
Title: Evaluation Of siMS Score As Amarker Of Metabolic Syndrome In Children With Simple Obesity
Brief Title: Metabolic Syndrome and Sims Score
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, BASMA SAYED, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: siMS SCORE
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Metabolic Syndrome , Sims Score and Pediatrics
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic Syndrome and Sims Score (Experimental)
  Interventions: Diagnostic Test: Sims Score

INTERVENTIONS:
Diagnostic Test: Sims Score — Evaluation Of siMS Score As Amarker Of Metabolic Syndrome In Children With Simple Obesity

SUMMARY:
SiMSscore was used as a simple and accurate method for Quantifying Metabolic Syndrome in adults , Developed siMS score was calculated using formula: siMS score = 2*Waist/Height + Gly/5.6 + Tg/1.7 + TAsystolic/130-HDL/1.02 or 1.28 (for male or female subjects, respectively),However studies on siMSscor in pediatric was done .

PsiMSscore(pediatric sims score) calculated using formula: (2xWaist/Height) + (Glucose(mmol/l)/5.6) + (triglycerides(mmol/l)/1.7) + (Systolic BP/130)-(HDL(mmol/l)/1.02(Soldatovic etal;2016).

DETAILED DESCRIPTION:
Metabolic Syndrome (MetS) is defined as a cluster of cardio metabolic risk factors that include central obesity low levels of high-density lipoprotein-cholesterol (HDL-C), hypertriglyceridemia, hypertension, and hyperglycaemia. Metabolic changes in childhood track into adulthood, predisposing these individuals to type 2 diabetes, and cardiovascular diseases.

The underlying prevalence of MetS in adolescents depends on the set of MetScri:eria used, with overall ranges in the US from 1.2%-9.8% using modified ATP-III criteria (Adult Treatment PanelII) to 4.5%-8.4% using the IDF adolescent criteria . Assessments among school-aged children and early adolescents islower (0.2%-1.2%) which is likely because of the strong effects of puberty on insulin resistance.

There is no consensus regarding the diagnosis of metabolic syndrome in children and adolescents. It is evident that each component of the syndrome must be identified as early as possible in order to prevent definitive lesion Pediatric and adolescent metabolic syndrome (MetS) criteria adapted from the National Cholesterol Education Program Adult Treatment Panel III (ATP lll),

1. Central Obesity (WC): WC ≥ 90th percentile .
2. High BP (mmHg) : Systolic or diastolic DBP≥ 90% for age, sex, height
3. High Triglycerides (mg/dL) : TG ≥ 110 mg/dL (≥1.24 mmol/L) .
4. HDL ≤ 40 mg/dL(<1.03 mmol/L).
5. High Fasting Glucose :≥100 mg/dL (5.6 mmol/L) or known T2DM. Individuals need to have at least three abnormalities in MetS components to be classified as havingMetS SiMSscore was used as a simple and accurate method for Quantifying Metabolic Syndrome in adults , Developed siMS score was calculated using formula: siMS score = 2*Waist/Height + Gly/5.6 + Tg/1.7 + TAsystolic/130-HDL/1.02 or 1.28 (for male or female subjects, respectively),However studies on siMSscor in pediatric was done .

PsiMSscore(pediatric sims score) calculated using formula: (2xWaist/Height) + (Glucose(mmol/l)/5.6) + (triglycerides(mmol/l)/1.7) + (Systolic BP/130)-(HDL(mmol/l)/1.02

ELIGIBILITY:
Inclusion Criteria:

* All obese patients aged from 7 to 17 years old.

Exclusion Criteria:

* All obesechildren

  * With endocrial and syndromatic obesity, (Endocrinal disease as hypothyroidism and Cushing's syndrome etc, syndromic obesity asPrader-Willi syndrome ,Alstrom-Hallgren syndrome, Bardet-Biedl syndrome, Beckwith-Wiedemansyndrome,etc…….)
  * Children on medications that affect lipid profile that include (β-Blockers ,Amiodarone ,Loop diuretics, Thiazide diuretics (high dose) ,Sodium-glucose co-transporter 2 (SGLT2) inhibitors ,Steroid Hormones/Anabolic Steroids, Antiviral Therapy ,Immunosuppressants ,Centrally Acting Medications as Anticonvulsants).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2020-12-29 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
sims score as screening method of metabolic syndrome in pediatric in one year | sims score as screening method of metabolic syndrome in pediatric in one year

CONTACTS AND LOCATIONS:
Overall Officials: noha gamal, professor, Study Director — Director
Locations (1):
- Assuit Univesrity, Asyut, Egypt